CLINICAL TRIAL: NCT00430365
Title: Relevance of Maintenance Therapy Using Lenalidomide (Revimid®) After Autologous Stem Cell Transplantation Patients Under the Age Of 65. (Open, Randomised, Multi-centric Trial Versus Placebo).
Brief Title: Maintenance Therapy Using Lenalidomide in Myeloma
Acronym: IFM2005-02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Intergroupe Francophone du Myelome (Network); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0400401; French PHRC (Other Grant/Funding Number: 0400401)
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Myeloma
Keywords: Myeloma; Revlimid; Maintenance therapy; Autologous Stem Cell Transplantation
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo group (Placebo Comparator): Administration of oral placebo
  Interventions: Drug: placebo
- lenalidomide group (Experimental): Administration of lenalidomide
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — oral drug
  Other Names: REVLIMID
  Arms: lenalidomide group
Drug: placebo — oral placebo
  Arms: placebo group

SUMMARY:
Maintenance treatment of myeloma.

ELIGIBILITY:
Inclusion Criteria:

* No signs of progression after transplant
* Effective contraception if necessary (oral contraception for females and barrier methods of contraception for sexually active males)
* No active severe infection
* Satisfactory restoration of the haematological parameters defined by: PN >1,000/mm3 and Platelets > 75,000/mm3
* Bilirubin < 35 umol/l and GOT/GPT/PAL<3N
* Creatinine < 160 umol/l.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 614 (Estimated)
Dates: Start 2006-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of Revlimid® at prolonging the duration of the post-transplant response. | 2 years

SECONDARY OUTCOMES:
Assess the impact of Revlimid® on the post-transplant complete response rate | 2 years
Compare survival without events and overall survival of patients in the lenalidomide arm with the control | 2 years
Evaluate the long-term tolerance of Revlimid® in post-transplant maintenance therapy. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: ATTAL Michel, Pr, Principal Investigator — University Hospital, Toulouse
Locations (77):
- Belgium (10):
  - ZNA Middelheim, Antwerp
  - Algemeen Centrumziekenhuis Antwerpen, Antwerp
  - UZA Antwerpen, Antwerp
  - Hôpital Saint Joseph, Arlon
  - Institut Jules Bordet, Brussels
  - UCL St Luc, Brussels
  - Hôpital Saint Joseph, Gilly
  - Hôpital Jolimont, Haine-Saint-Paul
  - Heilig Hart Ziekenhuis, Roeselare
  - UCL Mont-Godinne, Yvoir
- France (58):
  - CH, Aix-en-Provence
  - CHRU, Amiens
  - CHRU Hôpital du Bocage, Angers
  - Centre hospitalier Argenteuil Victor Dupouy, Argenteuil
  - Centre hospitalier Duffaut, Avignon
  - Centre hospitalier de la côte basque, Bayonne
  - Hôpital Jean Minjoz, Besançon
  - CH, Blois
  - Hôpital Avicenne, Bobigny
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CHRU Hôpital haut Lévêque, Bordeaux
  - Hôpial Morvan, Brest
  - Polyclinique du Parc, Caen
  - Centre Baclesse, Caen
  - CH, Chartres
  - CH William Morey, Châlon-sur-Saône
  - Hôpital Antoine Béclère, Clamart
  - Hôpital d'instruction des Armées Percy, Clamart
  - CHRU Hôtel Dieu, Clermont-Ferrand
  - CH Louis Pasteur, Colmar
  - CHU Henri Mondor, Créteil
  - CHRU Dijon, Dijon
  - Centre hospitalier général, Dunkirk
  - CHRU Hôpital Michallon, Grenoble
  - Centre hospitalier départemental, La Roche-sur-Yon
  - CH, Le Mans
  - CHRU Hôpital Claude Huriez, Lille
  - Centre hospitalier Bodelio, Lorient
  - Centre Léon Bérard, Lyon
  - CHU Hôpital Edouard Herriot, Lyon
  - Institut Paoli Calmette, Marseille
  - Hôpital Nord, Marseille
  - Hôpital Notre Dame de Bon Secours, Metz
  - CHRU Hôpitaux de Brabois, Nancy
  - CHRU Hôtel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hôpital Archet, Nice
  - Hôpital de l'Archet, Nice
  - Hôtel Dieu, Paris
  - Hôpital Cochin, Paris
  - CHU Hôpital St Antoine, Paris
  - Centre hospitalier Lyon Sud, Pierre-Bénite
  - CHRU Hôpital Jean Bernard, Poitiers
  - Centre hospitalier de la région d'Annecy, Pringy
  - Hôpital Debré, Reims
  - CHRU Hôpital de Pontchaillou, Rennes
  - CHRU Hôpital Sud, Rennes
  - Centre hospitalier de Roanne, Roanne
  - Centre Henri Becquerel, Rouen
  - Centre hospitalier Yves Le Foll, Saint-Brieuc
  - Centre hospitalier de la Réunion, Saint-Denis
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - CHRU Hôpital de Hautepierre, Strasbourg
  - CHU Toulouse Purpan, Toulouse
  - CHU Toulouse Rangueil, Toulouse
  - CHRU Hôpital Bretonneau, Tours
  - Centre hospitalier, Troyes
  - CH Chubert, Vannes
- Switzerland (9):
  - Center of Oncology/Hematology and transfusion Medicine, Kantonsspital, Aarau
  - Universitäts Spital, Basel
  - Istituto Oncologico Sviss. Italiana IOSI Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital, Bern
  - Hôpital cantonal, Genêve
  - CHUV, Lausanne
  - Onkologie/Hämatologie Kantonsspital st Gallen, Sankt Gallen
  - Spital Thun-Simmental Onkologiezentrum, Thun
  - Institute of Oncology and Hematology Stadtspital Triemli, Zurich

REFERENCES:
- [Background] Combination chemotherapy versus melphalan plus prednisone as treatment for multiple myeloma: an overview of 6,633 patients from 27 randomized trials. Myeloma Trialists' Collaborative Group. J Clin Oncol. 1998 Dec;16(12):3832-42. doi: 10.1200/JCO.1998.16.12.3832. PMID 9850028
- [Derived] Attal M, Lauwers-Cances V, Marit G, Caillot D, Moreau P, Facon T, Stoppa AM, Hulin C, Benboubker L, Garderet L, Decaux O, Leyvraz S, Vekemans MC, Voillat L, Michallet M, Pegourie B, Dumontet C, Roussel M, Leleu X, Mathiot C, Payen C, Avet-Loiseau H, Harousseau JL; IFM Investigators. Lenalidomide maintenance after stem-cell transplantation for multiple myeloma. N Engl J Med. 2012 May 10;366(19):1782-91. doi: 10.1056/NEJMoa1114138. PMID 22571202